CLINICAL TRIAL: NCT06737471
Title: Italian Cp eArly REhabilitation (iCARE)
Brief Title: Cp eArly REhabilitation
Acronym: iCARE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 1114
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: cerebral-palsy; children; pediatric; intervention; rehabilitation; motor; cognitive
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Extensive rehabilitation treatment: A 3-hour weekly rehabilitation treatment is delivered to each patient in an outpatient setting for 15 weeks.
  Interventions: Other: Extensive rehabilitation treatment
- Intensive rehabilitation treatment: A 3-hour daily rehabilitation treatment is delivered to each patient in the care units of the Hospital for 5 weeks.
  Interventions: Other: Intensive rehabilitation treatment

INTERVENTIONS:
Other: Intensive rehabilitation treatment — A 3-hour daily rehabilitation treatment will be delivered to each patient 5 days a week for 5 weeks (45 hours) in the care units of the Hospital.
  Rehabilitation will address the following macro goals: gross motor, manipulative, visual and visual-cognitive.
  Groups: Intensive rehabilitation treatment
Other: Extensive rehabilitation treatment — A 3-hour weekly rehabilitation treatment will be delivered to each patient for 15 weeks (45 hours) in an outpatient setting.
  Rehabilitation will address the following macro goals: gross motor, manipulative, visual and visual-cognitive.
  Groups: Extensive rehabilitation treatment

SUMMARY:
The present study aims to investigate the efficacy of play-based rehabilitation delivered as usual care in children with cerebral palsy in a rehabilitation center offering both intensive and extensive care. Up to now, few studies described and examined treatments' efficacy in this population.

Secondary aim of the study will be comparing the efficacy of the two rehabilitation treatment formats (intensive vs. extensive), which will have the same dose (sessions delivered) and ingredients (content). The intervention delivered as extensive care (3 sessions per week per 15 weeks) will be offered in community rehabilitation centers (Centri di Riabilitazione-CDR), while the one delivered as intensive care (3 sessions daily per 5 days a week for 3 weeks) will be offered to children admitted to hospital inpatient care units. This comparison allows verifying if delivery time may affect outcomes.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common cause of disability in childhood and is characterized by permanent disorders of movement and posture development, causing important limitations in autonomy. CP is attributable to non-progressive disorders that occur in the fetal and infant brain during development. Motor disorders are often accompanied by epilepsy, secondary musculoskeletal problems and impairments in different areas, such as sensory and perceptual domains, intelligence, communication abilities and behavior regulation.

The criteria for early diagnosis of CP have been refined over time and now it may be possible to obtain a diagnosis also when the child is less than 5 months of age, when movement alterations can be detected by clinicians and neuroradiological data may confirm the diagnosis, allowing early and ad hoc patients' management in an important period for brain plasticity. In the Italian context, delays in access and limitations in the continuity of care process have been found. After diagnosis, it is fundamental to use specific tools designed to assess and classify the severity of the CP. In the motor domain, the Gross Motor Function Classification System (GMFCS) and the Manual Ability Classification System (MACS) are used to examine for manipulative skill activities. Communication skills can be assessed by using the Communication Function Classification System, visual abilities by using the Visual Function Classification System (VFCS) and aspiration risk by using the Eating and Drinking Ability Classification System (EDACS). Cognitive aspects should be assessed by adopting the age-related Wechsler scales. When it is not possible to administer these scales, that is to children aged less than 2.5 years or to those presenting with aphasia, blindness, or severe cognitive difficulties, different tools should be used, such as the Griffiths Mental Development Scales (GMDS), measuring and assessing the developmental rates of children from birth to age 6. The combination of data based on these tools allows having an overall picture of the of child's functioning.

Early interventions are based on the following principles: (1) facilitating the child's active movements rather than focusing only on stretching or passive movements; (2) setting up an enriched play environment to increase stimulation and motivation; (3) improving developmental skills to favor developmental progress. Rehabilitation interventions delivered in accordance with these three principles should be guided by a pathology-specific assessment and aimed at addressing specific objectives and clearly measuring the results. Follow-up monitoring of the child is essential to assess the effectiveness of interventions and update treatment plans, by adapting interventions to the progressive needs of each child, which could optimize treatment outcomes. By adhering to evidence-based practices following the latest scientific evidence, healthcare professionals may enhance the quality of the care and, as a consequence, the likelihood of positive better quality of life for children. Nevertheless, up to now, few studies described and examined treatments' efficacy in this population focusing on the best format to adopt; also, no clear indications on whether a different setting (intensive vs extensive) for intervention delivery may lead to different outcomes are available.

With respect to the motor domain, it has been highlighted the importance to deliver interventions that favor the autonomous exploration of the environment by the child and include strategies to sustain purposeful movements. The evidence, although limited, seems to suggest that "movement tasks" that support the motivation of the child to try to complete an activity and to reach a goal, even through trial and error, should be used. In order to plan an intervention personalized for each child, it is essential to take into account the topographical characteristics of the motor impairment. Specific rehabilitation proposals for upper limb rehabilitation in the hemiplegic child have already been reported.

In line with the principles of a family-centered-care approach, clinicians should involve parents and caregivers in the care process, so that they may have an active role in the child's rehabilitation practice outside the clinic. In fact, parents may play a fundamental role in setting the goals of the therapy practice in the ecological setting and may choose tasks at an appropriate level of difficulty for their child. Further, they may to expose the child to enjoyable motor activities performed in an enriched environment with adequate frequency and intensity, so that new motor skills can be developed and learned. Rehabilitation approaches such as the 'Goals-Activity-Motor Enrichment' (GAME), based on the combination of motor training, interaction with the environment, environmental enrichment, and parental coaching, and the 'Small Step Program' [19], based on the promotion of gross-motor and postural skills, the use of hands for environmental exploration and communication, are clear examples of the implementation of the principles outlined above.

However, the literature on early interventions for high-risk infants is still at an embryonic phase: studies are heterogeneous, provide weak evidence on outcomes and their methodological quality is limited. Generally, for all neurological disabilities guidance on how to develop and deliver appropriate, targeted, and evidence-based rehabilitation interventions is limited. Therefore, it is necessary to conduct further research on the topic.

In many cases, the evidence of treatment response has not been robust enough to demonstrate a change in trained functions that is clinically, statistically, and economically important. In this regard, Rob Forsyth and colleagues have suggested that the exclusive focus on therapy dose could be misleading, as rehabilitation content should also be precisely captured.

In our Institute (Scientific Institute IRCCS E. Medea, Bosisio Parini, Lecco, Italy) rehabilitation interventions are delivered both in community rehabilitation centers (Centri di Riabilitazione-CDR), where activities are offered as extensive care, and in the inpatient care units of the Hospital, where shorter but more intensive rehabilitation interventions are offered. For both treatment delivery options, decades of experience have been collected. In this study, we aim at assessing the global efficacy of rehabilitation interventions offered as usual care, together with comparing the efficacy of intensive and extensive treatment formats . This is to evaluate if time and intensity in rehabilitation delivery can be considered a mediator variable affecting outcomes. Both interventions have the same treatment dose (sessions delivered) and ingredients (content).

ELIGIBILITY:
Inclusion Criteria:

* age between 6 months (corrected age in case of prematurity) and 5 years;
* a diagnosis of cerebral palsy due to perinatal suffering, neurological syndromes, rare diseases with neurological impairment or congenital diseases of unknown nature.

Exclusion Criteria:

* profound deafness and/or severe hypovisus/blindness;
* a diagnosis of neurodegenerative diseases, acquired brain injury or brain tumor.

Ages: 36 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy aged 6 months to 5 years receiving rehabilitation as usual care will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure for children (WeeFIM) | At baseline, immediately after the intervention and at an 8-month follow-up.
  The WeeFIM scale assesses the ability of a child in day-to-day functional tasks related to the 3 following main domains: self-care, mobility and cognition. It is composed of 18 items, each evaluating child's performance on a 7-point ordinal scale. WeeFIM is usually adopted in typically developing children aged 6 months-7 years. However, for children with developmental disabilities, the scale can be used up to 21 years.
The Gross Motor Function Measure 88 (GMFM-88) | At baseline, immediately after the intervention and at an 8-month follow-up.
  The Gross Motor Function Measure 88 (GMFM-88) allows measuring changes in gross motor function over time or with intervention in children with cerebral palsy. Items span the spectrum of gross motor activities in 5 dimensions 1) Lying and Rolling; 2) Sitting; 3) Crawling and Kneeling; 4) Standing; 5) Walking, Running and Jumping. Items evaluate performance on a 3-point Likert scale. Higher scores indicate better performance.

SECONDARY OUTCOMES:
The Behavior Rating Inventory of Executive Function-Preschool Version -parent form | At baseline, immediately after the intervention and at an 8-month follow-up.
  The Behavior Rating Inventory of Executive Function-Preschool Version -parent form is a parent report assessing specific components of executive functions through observable everyday behaviors in children aged 2 to 5:11 years. It has 5 clinical scales (Inhibit, Shift, Emotional Control, Working Memory, Plan/Organize), 3 composite indices (Inhibitory Self-Control Index (ISCI), Flexibility Index (FI), Emergent Metacognition Index (EMI)), and an overall composite score known as the Global Executive Composite (GEC).

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale Diurno, Como, Como
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale Diurno e Residenziale, Bosisio Parini, Lecco
  - Scientific IRCCS, E. Medea, Bosisio Parini, Lecco
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale, Sesto San Giovanni, Milano
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale, Carate Brianza, Monza E Brianza
  - Associazione "La Nostra Famiglia" - Centro di Riabilitazione Ambulatoriale Diurno, Vedano Olona, Varese

REFERENCES:
- [Background] Ko J, Kim M. Reliability and responsiveness of the gross motor function measure-88 in children with cerebral palsy. Phys Ther. 2013 Mar;93(3):393-400. doi: 10.2522/ptj.20110374. Epub 2012 Nov 8. PMID 23139425
- [Background] Duku E, Vaillancourt T. Validation of the BRIEF-P in a sample of Canadian preschool children. Child Neuropsychol. 2014;20(3):358-71. doi: 10.1080/09297049.2013.796919. Epub 2013 May 31. PMID 23721091
- [Background] Msall ME, DiGaudio K, Rogers BT, LaForest S, Catanzaro NL, Campbell J, Wilczenski F, Duffy LC. The Functional Independence Measure for Children (WeeFIM). Conceptual basis and pilot use in children with developmental disabilities. Clin Pediatr (Phila). 1994 Jul;33(7):421-30. doi: 10.1177/000992289403300708. PMID 7525140
- [Background] Morgan C, Fetters L, Adde L, Badawi N, Bancale A, Boyd RN, Chorna O, Cioni G, Damiano DL, Darrah J, de Vries LS, Dusing S, Einspieler C, Eliasson AC, Ferriero D, Fehlings D, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Mak C, Maitre N, McIntyre S, Mei C, Morgan A, Kakooza-Mwesige A, Romeo DM, Sanchez K, Spittle A, Shepherd R, Thornton M, Valentine J, Ward R, Whittingham K, Zamany A, Novak I. Early Intervention for Children Aged 0 to 2 Years With or at High Risk of Cerebral Palsy: International Clinical Practice Guideline Based on Systematic Reviews. JAMA Pediatr. 2021 Aug 1;175(8):846-858. doi: 10.1001/jamapediatrics.2021.0878. PMID 33999106
- [Background] Baranello G, Signorini S, Tinelli F, Guzzetta A, Pagliano E, Rossi A, Foscan M, Tramacere I, Romeo DMM, Ricci D; VFCS Study Group. Visual Function Classification System for children with cerebral palsy: development and validation. Dev Med Child Neurol. 2020 Jan;62(1):104-110. doi: 10.1111/dmcn.14270. Epub 2019 Jun 10. PMID 31180136
- [Background] Hidecker MJ, Paneth N, Rosenbaum PL, Kent RD, Lillie J, Eulenberg JB, Chester K Jr, Johnson B, Michalsen L, Evatt M, Taylor K. Developing and validating the Communication Function Classification System for individuals with cerebral palsy. Dev Med Child Neurol. 2011 Aug;53(8):704-10. doi: 10.1111/j.1469-8749.2011.03996.x. Epub 2011 Jun 27. PMID 21707596
- [Background] Novak I, Morgan C, Adde L, Blackman J, Boyd RN, Brunstrom-Hernandez J, Cioni G, Damiano D, Darrah J, Eliasson AC, de Vries LS, Einspieler C, Fahey M, Fehlings D, Ferriero DM, Fetters L, Fiori S, Forssberg H, Gordon AM, Greaves S, Guzzetta A, Hadders-Algra M, Harbourne R, Kakooza-Mwesige A, Karlsson P, Krumlinde-Sundholm L, Latal B, Loughran-Fowlds A, Maitre N, McIntyre S, Noritz G, Pennington L, Romeo DM, Shepherd R, Spittle AJ, Thornton M, Valentine J, Walker K, White R, Badawi N. Early, Accurate Diagnosis and Early Intervention in Cerebral Palsy: Advances in Diagnosis and Treatment. JAMA Pediatr. 2017 Sep 1;171(9):897-907. doi: 10.1001/jamapediatrics.2017.1689. PMID 28715518